CLINICAL TRIAL: NCT01168544
Title: Vitamin D Supplementation in Elderly Nursing Home Residents: Daily Supplementation Compared to a Loading Dose an Monthly Supplementation, a Randomised Trial
Brief Title: Daily Vitamin D Supplementation Compared to a Loading Dose and Monthly Supplementation in Elderly Nursing Home Residents
Acronym: VIDIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Mw. D.T.W. Salemink, Alysis Zorggroep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTC 712-050710
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Vitamin D Deficiency in Older Persons
Keywords: Vitamin D; Colecalciferol; Nursing home; Loading dose
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- loading dose and 50.000 IU vit D3/month (Experimental): Loading dose based on body weight and baseline serum 25 (OH)D level + 50.000 IU vit D3/month consolidation
  Interventions: Dietary Supplement: loading dose Vitamin D and 50.000 IU vit D3/month
- Loading dose and 25.000 IU vit D3/month (Experimental): Loading dose based on body weight and baseline serum 25(OH)D level + 25.000 IU vit D3/month consolidation therapy
  Interventions: Dietary Supplement: loading dose and 25.000 IU vit D3/month
- 800 IU vit D3/dag (Active Comparator): 800 IU vit D3/dag
  Interventions: Dietary Supplement: Vitamin D 800 IU /day

INTERVENTIONS:
Dietary Supplement: loading dose Vitamin D and 50.000 IU vit D3/month — loading dose based on body weight and baseline serum 25(OH)D level + 50.000 IU vit D3/month consolidation therapy
  Arms: loading dose and 50.000 IU vit D3/month
Dietary Supplement: loading dose and 25.000 IU vit D3/month — loading dose based on body weight and baseline serum 25(OH)D level + 25.000 IU vit D3/month consolidation therapy
  Arms: Loading dose and 25.000 IU vit D3/month
Dietary Supplement: Vitamin D 800 IU /day — 800 IU vit D3/day
  Arms: 800 IU vit D3/dag

SUMMARY:
Vitamin D deficiency is common in older persons, in particular in residents of nursing homes. This is mainly explained by the fact that older persons do not often go outside in the sunshine. On top of that the capacity of the skin to synthesize provitamin D is decreased and dietary vitamin D intake is low. Vitamin D deficiency leads to osteoporosis, falls and fractures. To prevent morbidity and mortality due to falls and fractures it seems logical to supplement vit D in order to correct the deficiency. The advised daily dose of vit D supplementation is 800 IU. Several studies showed that with this dose the required serum 25(OH)D levels will not be reached.

primary objective of this study is:

* to investigate whether with a loading dose based on body weight and baseline serum 25(OH)D level more patients reach adequate serum 25(OH)D levels compared to 800 IU a day.
* to determine the best consolidation treatment.

Secondary objective

* is a loading dose based on body weight and baseline serum 25(OH)D level safe to use in residents of nursing homes.
* is there a relation between the increase in serum 25(OH)D level and muscle strength (handgrip strength).
* is there a relation between the increase in serum 25(OH)D level and mobility (2 minute walk test).

Study design:

Randomised trial with 3 study groups:

* Group 1a. loading dose based on body weight and baseline serum 25(OH)D level + 50.000 IU vit D3/month consolidation therapy.
* Group 1b. loading dose based on body weight and baseline serum 25(OH)D level + 25.000 IU vit D3/month consolidation therapy.
* Group 2. 800 IU vit D3/ dag.

Study population:

Vitamine D deficient residents of nursing homes, 65 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Long term indication for living in a residential home for the elderly
* Age > 65 years
* Vitamin D deficiency (serum 25- hydroxycholecholecalciferol (25(OH)D3 < 50 nmol/l)
* Informed Consent

Exclusion Criteria:

* Hypercalcemia (serum CA > 2.60 mmol/l)
* Life expectancy < 1/2 year
* Multivitamin use including > 400 IE vit D
* Non-functional dominant arm

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-05

PRIMARY OUTCOMES:
Proportion of patients reaching an adequate serum 25(OH)D level (75-150 nmol/l)

SECONDARY OUTCOMES:
Proportion of patients reaching a serum 25(OH)D level > 220 nmol/l
Handgrip strength
Distance achieved in a 2 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: D.T.W. Salemink, Drs., Principal Investigator — Alysis Zorggroep
Locations (1):
- Alysis Zorggroep, verpleeghuis zevenaar, Zevenaar, Gelderland, Netherlands